CLINICAL TRIAL: NCT00652678
Title: Predictive Blood Tests for Severe Radiation Reactions in Breast Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Carol M. Baldwin Breast Cancer Research Fund, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Project # 1050425
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2013-09

CONDITIONS: Abnormalities, Radiation-Induced
Keywords: Breast cancer; Radiation effects
MeSH Terms: conditions — Abnormalities, Radiation-Induced; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Some patients who undergo breast cancer treatment with lumpectomy followed by radiation therapy develop significant late skin and soft tissue changes, resulting in a poor cosmetic outcome. The goal of this study is to try to predict severe tissue reactions by using a combination of three of the latest blood tests, one of which we have developed ourselves.

DETAILED DESCRIPTION:
Three tubes of blood will be drawn from each subject. Two members of the study team will also independently assess each subject for the degree to which various radiation-induced soft tissue changes are evident. Subjects will be put into three groups according to the severity of the soft tissue changes which are noted, and the results of the blood tests for members of each group will be analyzed to determine whether a correlation with cosmetic outcomes can be determined. If the results are promising, they will be studied further and used as the basis for future prospective clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer treatment: lumpectomy followed by external beam XRT to breast
* Age at the time of radiotherapy treatment: 45-65 years old
* XRT dose to breast: >/= 4500 and </= 5200 cGy, fraction size 180 or 200 cGy
* Dose distribution: no area receiving >/= 112% of prescribed dose
* Follow-ups: patients must be >/= 2.5 years post-treatment

Exclusion Criteria:

* Reconstructive surgery to involved breast

Min Age: 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be drawn from patients with a history of treatment for breast cancer with lumpectomy followed by radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
correlation of the results obtained from the three blood tests with the clinical assessments of cosmetic outcome for each subject | at least 2.5 years following lumpectomy and radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Hahn, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States